CLINICAL TRIAL: NCT02901496
Title: The Role of Exercise Training Combined With Tocilizumab on Visceral and Epicardial Adipose Tissue and Gastric Emptying in a High Risk Population: an Exploratory Double-blind, Placebo-controlled Randomised Trial
Brief Title: Ectopic Adipose Tissue, Exercise Training and IL-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Lang Lehrskov, MD, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-16018062
Record Dates: First submitted 2016-08-01; First posted 2016-09-15 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2022-06

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity | interventions — Resistance Training; tocilizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Endurance exercise + infusion of Tocilizumab (Experimental): Endurance exercise training + monthly infusion of Tocilizumab
  Interventions: Behavioral: Endurance Exercise Training; Drug: Tocilizumab
- Endurance exercise + infusion of placebo (Experimental): Endurance exercise training + monthly infusion of placebo
  Interventions: Behavioral: Endurance Exercise Training; Drug: Placebo
- No exercise + infusion of Tocilizumab (Experimental): No exercise + monthly infusion of Tocilizumab
  Interventions: Behavioral: No Exercise; Drug: Tocilizumab
- No exercise + infusion of placebo (Placebo Comparator): No exercise training + monthly infusion of placebo
  Interventions: Behavioral: No Exercise; Drug: Placebo
- Resistance exercise + infusion of placebo (Experimental): Resistance exercise training + monthly infusion of placebo
  Interventions: Behavioral: Resistance Exercise Training; Drug: Placebo

INTERVENTIONS:
Behavioral: Endurance Exercise Training — Three months of supervised training. Interval training, 3 sessions weekly of 45 min. During intervals the intensity will be minimum 70 % of VO2 max
  Other Names: Endurance exercise
  Arms: Endurance exercise + infusion of Tocilizumab; Endurance exercise + infusion of placebo
Behavioral: Resistance Exercise Training — Three months of supervised resistance training. Subjects will perform 3 weekly sessions of 45 min. The intensity will be kept at minimum 60% of 1RM.
  Other Names: Resistance exercise
  Arms: Resistance exercise + infusion of placebo
Behavioral: No Exercise — Control to exercise
  Arms: No exercise + infusion of Tocilizumab; No exercise + infusion of placebo
Drug: Tocilizumab — Tocilizumab infusion will be administered monthly (8 mg/kg body weight i.v., maximun 800 mg). Each subject will receive 3 infusions during the study period.
  Other Names: RoActemra
  Arms: Endurance exercise + infusion of Tocilizumab; No exercise + infusion of Tocilizumab
Drug: Placebo — Saline infusion will be administered monthly (same volume as Tocilizumab). Each subject will receive 3 infusions during the study period.
  Other Names: Saline
  Arms: Endurance exercise + infusion of placebo; No exercise + infusion of placebo; Resistance exercise + infusion of placebo

SUMMARY:
Aim: Exercise training improves the risk of cardiometabolic diseases; yet the underlying mechanisms are unclear. Exercise induces release of IL-6 from skeletal muscle. Acute elevations in IL-6 improve lipid and glucose metabolism, the latter partly through a delayed gastric emptying. Physical inactivity causes accumulation of visceral fat (VAT). Visceral and epicardial adipose tissue (EAT) is more inflamed than subcutaneous adipose tissue. Thus, the investigators hypothesize that exercise-induced IL-6 mediates the exercise-induced reduction in EAT and VAT. Secondly, the investigators hypothesize that exercise-induced adaptations in glucose metabolism and gastric motility are dependent on IL-6. Finally the investigators hypothesise that both endurance and resistance exercise training reduce VAT and EAT.

Primary aim: To investigate the effects of exercise training on VAT and to determine to what extend IL-6 mediates this effect.

Secondary aims: 1) To determine whether 12 weeks of endurance and strength training can reduce the amount of EAT. 2) To study whether the effects of exercise on glucose metabolism and gastric emptying are dependent on IL-6.

Methods: Inclusion: 70 inactive men and women, >18 years, waist to height ratio > 0.5 and/or waist circumference ≥ 88 cm (women); waist circumference ≥ 102 cm (men) Design: A 12-week, double-blinded randomised, placebo-controlled exercise intervention study.

Intervention: Subjects will be randomised to one of five groups: i) Tocilizumab (IL-6 receptor antibody) and endurance training, ii) Placebo to Tocilizumab and endurance training, iii) Tocilizumab, no exercise iv) Placebo to Tocilizumab and no training, and v) Placebo to Tocilizumab, and resistance training. Tocilizumab/placebo dose will be administered (according to standard recommendations) before the first training session, and maintained during the 12-week training program. Training will be supervised to ensure intensity and compliance. Subjects will be instructed not to change eating habits and informed that this study does not aim for a weight loss.

Statistical considerations: Study investigators are blinded to treatment allocation. Dropouts will be replaced. A sample size of 70 subjects is needed to detect a 10% change in visceral adipose, with a power of 80% and a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Sedentary
* Waist to height ratio ≥ ½ and/or waist circumference ≥ 88 cm (women); waist circumference ≥ 102 cm (men)
* Age ≥ 18 y

Exclusion Criteria:

* Pregnancy
* Diagnosed with diabetes (HbA1c ≥ 48 mmol/mol or fasting glucose ≥ 7.0 mmol/l)
* Diagnosed with ischemic heart disease
* Atrial fibrillation
* Treatment with biologic rheumatic drugs, systemic prednisolone or other immunosuppressive treatments
* Health conditions that prevents individuals from participating in the exercise training intervention e.g. severe obesity
* Patients who cannot undergo MRI scans (e.g. kidney disease, metallic implants or claustrophobia)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Changes in visceral fat mass | 0, 12 weeks
  Visceral fat mass will be measured by MRI before and after the intervention. Difference in change in visceral fat mass from baseline to 12 weeks follow up will be compared between group: Endurancetraining + tocilizumab and group: Endurancetraining + placebo.

SECONDARY OUTCOMES:
Changes in visceral fat mass | 0, 12 weeks
  Difference in change in visceral fat mass from baseline to 12 weeks follow up will be compared between group: Endurancetraining + placebo and group: no training + placebo.
Changes in visceral fat mass | 0, 12 weeks
  2. Difference in change in visceral fat mass from baseline to 12 weeks follow up will be compared between group: Endurancetraining + placebo and group: resistance training + placebo.
Changes in visceral fat mass | 0, 12 weeks
  3. Difference in change in visceral fat mass from baseline to 12 weeks follow up will be compared between group: Endurancetraining + tocilizumab and group: no training + tocilizumab.
Changes in visceral fat mass | 0, 12 weeks
  4. Difference in change in visceral fat mass from baseline to 12 weeks follow up will be compared between group: resistance training + placebo and group: no training + placebo.
Changes in visceral fat mass | 0, 12 weeks
  5. Difference in change in visceral fat mass from baseline to 12 weeks follow up will be compared between group: no training + placebo and group: no training + tocilizumab.
Epicardial adipose tissue | 0, 12 weeks
  Cardiac fat volume will be measured by a cardiac MRI scan before and after the interventions. All groups will be compared.
Gastric emptying | 0, 12 weeks
  Gastric emptying will be measured by paracetamol blood levels (mmol/l) before and after the interventions.
  The paracetamol levels will be compared between groups as follows. Group: Endurancetraining + tocilizumab and group: Endurancetraining + placebo. Group: Endurancetraining + placebo and group: no training + placebo. Group: Endurancetraining + tocilizumab and group: no training + tocilizumab. Group: No training + placebo and group: no training + tocilizumab.

OTHER OUTCOMES:
Peri- and paracardial adipose tissue volume (measured by MRI) | 0, 12 weeks
Body composition analysis (measured by Dual-energy X-ray absorptiometry) | 0, 4, 8 and 12 weeks
Waist circumference (measured in cm) | 0, 4, 8 and 12 weeks
BMI (kg/m^2, weight in kilograms, height in meters) | 0, 4, 8 and 12 weeks
Resting blood pressure as a measure of cardiovascular function | 0, 12 weeks
Maximal aerobic capacity (cardiovascular fitness) (VO2 peak) | 0, 12 weeks
Muscle strength measured by one repetition maximum (1RM) | 0, 12 weeks
Oral glucose tolerance test | 0, 12 weeks
Glycemic control during mixed meal tolerance test | 0, 12 weeks
Free-living glycemic control using continuous glucose monitoring | 0, 12 weeks
Pro- and anti-inflammatory cytokines(Interleukin-6, Interleukin-1ra, Interleukin-1, Interleukin-18, Interleukin-15, Interleukin-10) | 0,4, 8 and 12 weeks
soluble Interleukin-6 receptor (sIL-6R) | 0,4, 8 and 12 weeks
soluble gp130 | 0,4, 8 and 12 weeks
Adipose characteristic by blood markers | 0,4, 8 and 12 weeks
  Blood sampling
Cortisol | 0,4, 8 and 12 weeks
  Blood sampling
Catecholamines (Epinephrine and norepinephrine) | 0,4, 8 and 12 weeks
leukocytes | 0,4, 8 and 12 weeks, (Timepoints: 0, 22, 45, 01:45, 02:45, at week 0 and 12)
  Blood sampling
Glucagon | 0,4, 8 and 12 weeks
  blood sampling
Blood lipid | 0,4, 8 and 12 weeks
  Blood sampling
Cardiovascular function assessed by blood markers | 0,4, 8 and 12 weeks
Inflammation status assessed by blood markers | 0,4, 8 and 12 weeks
Adipose biopsy to assess the adipokine expression signature | 0, 12 weeks
Photo of subjects | 0, 12 weeks
  To asses if the visual appearance of the stomach is reflecting the amount of visceral fat mass and to see if there is a difference in the visual appearance before and after the intervention
Faecal and urine samples to asses changes in the microbiome | 0, 12 weeks
Change in sleepiness | 0, 12 weeks
  Self-report using the Epworth questionnaire
Exercise factors during an acute exercise bout | Timepoints: 0, 22, 45, 01:45, 02:45, before and after the intervention (0,12 weeks)
  cortisol, il-6, epinephrine and norepinephrine
Glucose metabolism during an acute exercise bout | Timepoints: 0, 22, 45, 01:45, 02:45, before and after the intervention (0,12 weeks)
  At each timepoint exercise factors: cortisol, il-6, epinephrine and norepinephrine will be measured. Furthermore pro anti-inflammatory cytokines, glucose, insulin, C-peptide, C-reactive protein will be reported.
Whole blood stimulation with Lipopolysaccharide and phytohaemagglutinin | During the acute exercise bout at Timepoints: 0, 22, 45, 01:45, 02:45, before and after the intervention (0,12 weeks)
  in vitro stimulation of whole blood.
Fibroblast growth factor 21 | During the acute exercise bout at Timepoints: 0, 22, 45, 01:45, 02:45, before and after the intervention (0,12 weeks)
oxidative burst in neutrophils | During the acute exercise bout at Timepoints: 0, 22, 45, 01:45, 02:45, before and after the intervention (0,12 weeks)
gastrointestinal health | 0,12 weeks
  A questionnaire regarding gastrointestinal symptoms. A Visual Analog Score will be used.
Physical activity | 0 weeks
  Self-report physical activity using The Minnesota Leisure Time Physical Activity Questionnaire
Diet registration | 0,4,12
  Self-report diet registration for 3 days
Satiety | 0,12
  self-report using a satiety questionnaire during mixed meal tolerance test
Cardiac function measured by heart rate recovery | 0, 12 weeks
Muscle biopsy to assess expression of exercise induced cytokines | 0, 12 weeks
Coronary sinus flow reserve as a measure of global perfusion using MRI | 0, 12 weeks
Insulin during mixed meal tolerance test | Time Frame: 0, 12 weeks
C-peptide during mixed meal tolerance test | Time Frame: 0, 12 weeks
Glucagon during mixed meal tolerance test | Time Frame: 0, 12 weeks
GLP-1 during mixed meal tolerance test | Time Frame: 0, 12 weeks
Insulin sensitivity index (Matsuda) based on mixed meal tolerance test | Time Frame: 0, 12 weeks
Insulin secretion index based on mixed meal tolerance test | Time Frame: 0, 12 weeks
IL-6 released in respons to an exercise bout | one of the first 3 and one of the last 3 exercise bouts
  IL-6 in plasma measured before and after an exercise bout

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, Professor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Centre of Inflammation and Metabolism (CIM) Centre for Physical Activity Research (CFAS), Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wedell-Neergaard AS, Lang Lehrskov L, Christensen RH, Legaard GE, Dorph E, Larsen MK, Launbo N, Fagerlind SR, Seide SK, Nymand S, Ball M, Vinum N, Dahl CN, Henneberg M, Ried-Larsen M, Nybing JD, Christensen R, Rosenmeier JB, Karstoft K, Pedersen BK, Ellingsgaard H, Krogh-Madsen R. Exercise-Induced Changes in Visceral Adipose Tissue Mass Are Regulated by IL-6 Signaling: A Randomized Controlled Trial. Cell Metab. 2019 Apr 2;29(4):844-855.e3. doi: 10.1016/j.cmet.2018.12.007. Epub 2018 Dec 27. PMID 30595477
- [Derived] Christensen RH, Wedell-Neergaard AS, Lehrskov LL, Legaard GE, Dorph E, Larsen MK, Launbo N, Fagerlind SR, Seide SK, Nymand S, Ball M, Vinum NB, Dahl CN, Henneberg M, Ried-Larsen M, Boesen MP, Christensen R, Karstoft K, Krogh-Madsen R, Rosenmeier JB, Pedersen BK, Ellingsgaard H. Effect of Aerobic and Resistance Exercise on Cardiac Adipose Tissues: Secondary Analyses From a Randomized Clinical Trial. JAMA Cardiol. 2019 Aug 1;4(8):778-787. doi: 10.1001/jamacardio.2019.2074. PMID 31268469
- [Derived] Christensen RH, Wedell-Neergaard AS, Lehrskov LL, Legard GE, Dorph EB, Nymand S, Ball MK, Zacho M, Christensen R, Ellingsgaard H, Rosenmeier JB, Krogh-Madsen R, Pedersen BK, Karstoft K. The role of exercise combined with tocilizumab in visceral and epicardial adipose tissue and gastric emptying rate in abdominally obese participants: protocol for a randomised controlled trial. Trials. 2018 May 2;19(1):266. doi: 10.1186/s13063-018-2637-0. PMID 29720225